CLINICAL TRIAL: NCT06249841
Title: Feasibility of in Vivo Percutaneous Cryobiopsy from the Human Bile Duct - CRYLEO
Brief Title: Feasibility of Cryobiopsy from the Bile Duct - CRYLEO
Acronym: CRYLEO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erbe Elektromedizin GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CIV-23-06-043299
Record Dates: First submitted 2024-01-05; First posted 2024-02-08 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Neoplasms, Bile Duct
MeSH Terms: conditions — Bile Duct Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Forceps biopsy against Cryoprobe biopsy (Experimental): A total of 6 forceps biopsies and 3 cryobiopsies will be taken for each patient, corresponding to a 2:1 ratio. The biopsies are divided into blocks of two (6 forceps, 3 cryo). The biopsy technique blocks are randomized, resulting in a sequence of 6 forceps biopsies followed by 3 cryobiopsies
  Interventions: Device: 1.1mm flexible Cryoprobe SU
- Cryoprobe biopsy against Forceps biopsy (Active Comparator): A total of 6 forceps biopsies and 3 cryobiopsies will be taken for each patient, corresponding to a 2:1 ratio. The biopsies are divided into blocks of two (6 forceps, 3 cryo). The biopsy technique blocks are randomized, resulting in a sequence of 3 cryobiopsies followed by 6 forceps biopsies.
  Interventions: Device: 1.1mm flexible Cryoprobe SU

INTERVENTIONS:
Device: 1.1mm flexible Cryoprobe SU — Six tissue samples retrieved by standard biopsy forceps and three samples by cryobiopsy (randomized sequence)
  Other Names: Comparator: SpyBite Max Forceps

SUMMARY:
This is a multi-center, prospective, feasibility study using a 1.1 mm flexible cryoprobe SU via percutaneous access in the bile duct. The device has a CE-approval. First feasibility and safety for application assessed in the bile duct performed ex vivo and in a patient case report study. The study will take place at 5 different sites in Germany. Recruitment is competitive. In total, 15 patients will be enrolled. Patients are screened for study inclusion at the participating hospitals.

Primary objective:

• Feasibility of percutaneous cryobiopsy in the bile duct

Secondary objectives:

* Size of biopsy (mean area (in mm2) of each biopsy technique)
* Percentage of successful retrievals of biopsies by each biopsy technique
* Representativeness of each biopsy sample
* Quality of each biopsy sample
* Grade of crash artifacts occurrence defined as crush artifact area per biopsy
* Rate of safety-relevant aspects, like for example bleeding, post-bleeding, perforation, infection and abscess

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of any neoplastic alterations in the bile duct system or other indication for biopsy sampling in the bile duct
* A percutaneous drainage or an access by means of percutaneous transhepatic cholangiodrainage (PTCD) has been previously established independent from study participation, without adverse events
* Patient is at least 18 years of age
* According to physicians' assessment, patient is able to follow study protocol or is able to understand the nature, objectives, benefits, implications, risks and inconveniences of the clinical investigation, able to comply with study requirements and understand and independently sign the Informed Consent Form

Exclusion Criteria:

* • Presence of hereditary bleeding disorder, e.g. hemophilia A or hemophilia B

  * Severe impairment of partial thromboplastin time (PTT) of >80s; International normalized ratio (INR) >3; platelet count <50,000 /nl
  * Dual antiplatelet therapy (change to aspirin monotherapy is no exclusion criterion)
  * Current use of systemic anticoagulation or antiplatelet therapy without the ability to hold therapy for the recommended amount of time prior to an invasive procedure (aspirin monotherapy is no exclusion criterion) Patient is participating in another clinical study pregnant or breast-feeding or intending to get pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study is feasibility of percutaneous cryobiopsy in the bile duct, i.e., successful retrieval of at least one cryobiopsy specimen per patient. | 30 days
  Feasibility of percutaneous cryobiopsy in the bile duct, i.e., successful retrieval of at least one cryobiopsy specimen per patient

SECONDARY OUTCOMES:
Size of biopsy (mean area (in mm2) of each biopsy technique) | 30 days
  Quality of biopsies
Percentage of successful retrievals of biopsies by each biopsy technique | 30 days
  Quality of biopsies
Representativeness of each biopsy sample | 30 days
  yes: evaluable bile duct epithelia in sufficient quantity and quality to make a diagnosis or no: absent or not sufficiently evaluable bile duct epithelia (e.g. crush artefacts, dissolved tissue association
Quality of each biopsy sample | 30 days
  Biopsy quality using a Likert-Scale for each biopsy technique
Grade of crash artifacts occurrence defined as crush artifact area per biopsy | 30 days
  Quality of biopsies
Rate of safety-relevant aspects, like for example bleeding, post-bleeding, perforation, infection and abscess | 30 days
  Quality of biopsies

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (5):
  - Klinikum Hamburg, Hamburg, Hamburg
  - Klinikum Hanau, Hanau, Hanau
  - Klinikum Essen, Essen, Hesse
  - Klinikum Nürnberg, Nuremberg, Nürnberg
  - Klinikum Stuttgart, Stuttgart, Stuttgart

REFERENCES:
- [Background] Peveling-Oberhag J, Zimmermann C, Linzenbold W, Ott G, Enderle M, Albert JG. Bile duct tissue acquisition by cholangioscopy-guided cryobiopsy technique: first-in-human application. VideoGIE. 2023 Feb 15;8(4):158-161. doi: 10.1016/j.vgie.2022.12.007. eCollection 2023 Apr. PMID 37095838
- [Background] Walter D, Peveling-Oberhag J, Schulze F, Bon D, Zeuzem S, Friedrich-Rust M, Albert JG. Intraductal biopsies in indeterminate biliary stricture: Evaluation of histopathological criteria in fluoroscopy- vs. cholangioscopy guided technique. Dig Liver Dis. 2016 Jul;48(7):765-70. doi: 10.1016/j.dld.2016.03.013. Epub 2016 Mar 26. PMID 27067926